CLINICAL TRIAL: NCT06682208
Title: Prospective Randomized Trial of Efficacy and Safety of Erector Spinae Catheter and Intercostal Nerve Cryoablation Protocols After Pectus Surgery
Brief Title: ES Catheter vs Cryoablation After Pectus Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-0760
Record Dates: First submitted 2024-11-07; First posted 2024-11-12 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Pectus Excavatum
MeSH Terms: conditions — Funnel Chest

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ES Catheter (Active Comparator): Hospital procedure for ES catheters will be followed for postoperative pain.
  Interventions: Procedure: ES catheter
- Intercostal Nerve Cryoablation (INC) (Active Comparator): Hospital procedure for intercostal nerve cryoablation will be followed for postoperative pain.
  Interventions: Procedure: Intercostal nerve cryoablation (INC)

INTERVENTIONS:
Procedure: ES catheter — ES catheter for postoperative pain control
  Arms: ES Catheter
Procedure: Intercostal nerve cryoablation (INC) — INC used for postoperative pain control
  Arms: Intercostal Nerve Cryoablation (INC)

SUMMARY:
Participants will be randomized to receive ES catheter or cryoablation for pain management after the Nuss procedure. The goal of this study is to compare the following between the two groups:

* Time to achieve short-term physical therapy goals and long-term functional outcomes
* Compare immediate and long-term postoperative opioid use
* Compare numbness on chest of postoperative day 1 and the return of sensation to baseline
* Compare the incidence of neuropathic pain and other complications

Participants will receive surveys for up to 12 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Age 12 - 21 years
* History of pectus excavatum
* Scheduled for Nuss procedure

Exclusion Criteria:

* Prior pectus repair
* Other concomitant surgeries
* Chronic pain conditions including Ehlers Danlos Syndrome
* Non-English speaking - rationale: the questionnaires used in the study are in English language and the social and cultural factors of pain perception of non-English speaking patients could affect the study power
* Severe developmental delays including cognitive (difficulties understanding), motor (cerebral palsy or muscular dystrophy), and speech delays (difficulties communicating)
* History of or active renal or liver disease
* Major surgery requiring opioids in the last 2 years
* Severe respiratory problems (such as obstructive sleep apnea, cystic fibrosis, pulmonary fibrosis, or pneumonia within the last month)
* Cardiac conditions including, but not limited to, cyanotic heart disease, hypoplastic left ventricle, arrhythmia, uncontrolled hypertension with ongoing treatment, Kawasaki disease, or cardiomyopathies. Participants with asymptomatic valvular lesions or defects may be included
* BMI >35
* Pregnant or breastfeeding females

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 176 (Estimated)
Dates: Start 2024-04-08 (Actual); Primary Completion 2029-04 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Compare time to reach discharge | Day of surgery up tp 10 days post-operative
  Comparing physical therapy goals to meet discharge criteria.

SECONDARY OUTCOMES:
Opioid consumption | Day of surgery to up to one year
  Comparing opioid consumption
Numbness on chest | Day of surgery and post-operative day 1
  An exam glove with ice will used on the anterior axillary line to obtain a rating of the sensation felt.
  0 - no sensation
  1. - lessened sensation
  2. - abnormal/painful sensation
  3. - no sensation
Neuropathic pain | Pre-operative, 6 weeks, 2-3 months, 4-6 months and 10-12 months post-operatively
  Surveys will be used to compare the incidence of neuropathic pain

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Walter, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Surya Narayanasamy, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States